CLINICAL TRIAL: NCT00759616
Title: Outcome Analysis of the Oxford Partial Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Dartmouth General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMET CA 03
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Knee Arthroplasty
Keywords: Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Oxford Partial Knee

INTERVENTIONS:
Device: Oxford Partial Knee — Oxford Partial Knee

SUMMARY:
Prospectively monitor the patients receiving the Oxford Partial knee arthroplasty

DETAILED DESCRIPTION:
Utilization of systematic outcome measurements and specific designated time frames to monitor patient satisfactions will assist in analysing this type of prosthesis and the post operative period. Data collected will be added to the compiled information from previous studies in relation to the Oxford knee.

ELIGIBILITY:
Inclusion Criteria:

* Patient Suitable for Knee Replacement

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2003-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
WOMAC, SF12, oxford Knee,KSCRS | 3weeks, 3months,6months, yearly

SECONDARY OUTCOMES:
Length of Hospital Stay | Postop

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth General Hospital, Dartmouth, Canada